CLINICAL TRIAL: NCT04179266
Title: Proof of Concept Study for Evaluation of the Effect of Ketamine Intranasal Spray in Treatment of Chronic Cluster Headache
Brief Title: Effect of Ketamine Intranasal Spray in Treatment of Chronic Cluster Headache
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CCH Pharmaceuticals (Industry)
Collaborators: Danish Headache Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001260-29
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: open label - proof of concept study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ketamine — One Cluster headache attack is treated with intranasal ketamine

SUMMARY:
Ketamine has been used clinically IV in a very safe manner by a very small number of clinicians, to treat migraines and CH, and various other rarer pain disorders, including mixed headache and neuropathic pain clinical syndromes. In 5 cases taken from Krusz J.C. headache clinic data in Dallas, Texas US, an intranasal spray of ketamine aqueous solution of 100 µL in one nostril were dosed in treatment of patients with refractory chronic cluster headache as an alternative to IV-treatment (data not published).The net conclusion, at this point, is that intranasal ketamine is a legitimate pharmacologic treatment and is safe and has in one case series proven effective for CH rescue.

The CCH patients will be dosed with an intranasal spray containing 172.5 mg ketamine hydrochloride (150 mg ketamine base) per ml in an aqueous solution. The individual dosing includes 15 mg ketamine in an intranasal sprayed volume of 100 µL given in one nose nostril under supervision of a nurse. The treatment is initiated at T0 under a CH attack when the headache pain exceeds NRS = 6 on an NRS pain scale. The first intranasal dose of 15 mg is given at time 0 and at time intervals of 6 minutes. At 15 minutes after 3 doses (45 mg) it is decided to evaluate whether the patient is sufficiently pain relieved (e.g. NRS < 4) or wants to receive rescue medications instead or if pain is not sufficiently relieved wants to continue until 5 dosing's (75 mg) are received at timepoints T24. The final evaluation of the treatment is performed at T30. Participants are followed up after 1-2 weeks by telehone

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between 18 and 60 years
* Diagnose: Chronic cluster headache according to ICHD-3 criteria (1)
* Body weight ≥50 kg and BMI ≤30

Exclusion Criteria:

* Conditions that result in the participant being unable to complete the experiment
* Medical history with elevated intraocular pressure (e.g. glaucoma)
* Medical history with severe heart or liver disease
* Aneurysmal vascular disease or arteriovenous malformations
* Medical history with severe neurological disease except of headache
* BP measured at baseline before CH attack (Systolic> 140 mmHg or / and diastolic blood pressure> 90 mm Hg)
* Medical history with severe depression or psychosis
* A previous history of drug abuse
* Consumption of illegal drugs within the last 6 months
* Medical history of nasal abnormality or dysfunction (e.g. rhinitis)
* High disposition for larynges or apnea
* Positive pregnancy test before treatment and breastfeeding
* Known hypersensitivity to ketamine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Effect on pain intensity at 15 min (50% reduction) | 15 minutes
  A 50% or more reduction in pain on a ten-point NRS scale (0: no pain, 10: worst imaginable pain) at T15 from pain intensity at T=0 .

SECONDARY OUTCOMES:
Effect on pain intensity at 30 min | 30 minutes
  A 50% or more reduction in pain on a ten-point NRS scale (0: no pain, 10: worst imaginable pain) at T30 from pain intensity at T=0.
Effect on pain intensity at 15 min (25% reduction) | 15 minutes
  A 25% reduction in pain on a ten-point NRS scale (0: no pain, 10: worst imaginable in) at T15 from pain intensity at T=0.
Proportion of patients achieving NRS less than 4 at 15 minutes | 15 minutes
  Proportion of patients achieving NRS less than 4 at 15 minutes
Proportion of patients achieving NRS less than 4 at 30 minutes | 30 minutes
  Proportion of patients achieving NRS less than 4 at 30 minutes
Proportion of patients receiving rescue medication at 15 minutes | 15 minutes
  Proportion of patients receiving rescue medication at 15 minutes
Proportion of patients preferring ketamine treatment compared to oxygen or injectable sumatriptan. | 180 minutes (entire attack)
  Proportion of patients preferring ketamine treatment compared to oxygen or injectable sumatriptan.
Proportion of patients experiencing serious side effects during treatment | one week follow-up.
  Proportion of patients experiencing serious side effects during treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No
Do to GDPR rules individual data will not be shared. Group data will be presented in publication. By request by other researcher other data will be presented if the request lines within the out approval from the The Danish Data Protection Agency